





**Pe**rsonalised **R**isk assessment in **F**ebrile illness to **O**ptimise **R**eal-life **M**anagement across the European Union (PERFORM)

| | | Chief investigator: Prof. Mike Principal Investigator: xxxxxxxxx | | |
|---|---|---|---|---|
| number: | | | rimcipai nivestigator. | ***** |
| | Consen | t form for children – pa | rents and guardi | ans to s |
| | | | | Please<br>initial if y<br>agree |
| 1. | I confirm that I have read and understand the information sheet version 1 dated 3 June 2016 for the above study and been given a copy to keep. I have had the opportunity to ask questions and have had these answered satisfactorily. | | | |
| 2. | I understand that participation is voluntary, and that I am free to withdraw consent from the study including the use of my child's samples and data at any time, without giving any reason and without my child's medical care or legal rights being affected | | | |
| 3. | I understand that sections of any of my child's hospital notes and data collected during the study may be looked at by responsible individuals from (local site name) or from regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to access my child's records. | | | |
| 4 | I agree to the use of my child's blood, DNA, nasal/throat swabs, urine and stool samples in this research project, as described on the patient information sheet. | | | |
| 5. | I agree for my child to take part in this research study | | | |
| 6. | I agree to the use of my child's samples in any future ethically-approved studies (this is optional). | | | |
| Name of Subject | | Signature (if able) | Date | |
| Name of Person taking consent | | Signature | Date | |



1 copy for subject; 1 copy for Principal Investigator; 1 copy to be kept with hospital notes.